CLINICAL TRIAL: NCT06141915
Title: Aerobic Training Combined With Diet Protocol on Immune System in Burn Patients.
Brief Title: Aerobic Training and Diet Protocol on Immune System in Burn Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Gamal Fawzy El-Sayed, Lecturer of physical therapy of surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004579
Record Dates: First submitted 2023-11-14; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Immune System Disorder
MeSH Terms: conditions — Immune System Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic training and diet protocol group (Experimental): 30 patients received aerobic training and diet protocol for 12 weeks.
  Interventions: Other: Aerobic training
- Aerobic training group (Experimental): 30 patients will receive aerobic training for 30 minutes, three times per week for 12 weeks.
  Interventions: Other: Aerobic training
- Diet protocol group (Active Comparator): 30 patients will receive diet protocol for 12 weeks.
  Interventions: Other: diet protocol

INTERVENTIONS:
Other: Aerobic training — patients will be engaged in aerobic training using treadmill three times per week, for 12 weeks. The exercise intensity will be 50-70% of each patient's maximum heart rate. Each exercise session will consist of three phases; five-minutes warming up phase in form of stretching exercises and walking on the treadmill at the slowest speed, 20-minutes conditioning phase in form of walking on the treadmill at 50% of participants' maximum heart rate in the first two weeks then progressed gradually to reach the 70% of maximum heart rate by the 12th weeks", and five-minutes cool down phase that will be constant as warming up phase. During the training, the patient's blood pressure, heart rate, and breathing pattern will be frequently monitored
  Arms: Aerobic training and diet protocol group; Aerobic training group
Other: diet protocol — diet protocol
  Arms: Diet protocol group

SUMMARY:
Aerobic exercises can produce immediate and short-term improvements in the immune response of leukocytes, T-lymphocytes, lymphocyte subpopulations, interleukins, and immunoglobulins. Even only a single session of aerobic exercises produces improvements in the utmost immune markers, such as T-lymphocytes, leukocytes, and immunoglobulins.

Also, burned patients suffer from post-traumatic stress and stress can cause this alteration through its effect on increasing the amounts of serum corticosteroid and catecholamine hormones, thus a decrease in the immunity response might occur. Increasing the aerobic capacity can significantly improve the mood. This might be attributed to the effect of aerobic exercises on decreasing stress hormones, like corticosteroids and catecholamines hormones.

The altered metabolism post major burn also affects the immune system in burn patients and the aerobic training enhances the metabolism, body composition and the lean mass and so, enhances the immune system.

One of the most important factors for a good and effective immune system is the balanced diet especially diet rich in vitamin D, fibers, and multiple nuts and seeds such as almond, walnut, pistachio, sunflower seeds, flax seeds and sesame seed that have an crucial role in improving the immune system either acting on it directly or indirectly by enhancing the general heath of the body and the patients mood.

DETAILED DESCRIPTION:
Group A (Aerobic training and diet protocol group): patients will be engaged in aerobic training using treadmill three times per week, for 12 weeks. The exercise intensity will be 50-70% of each patient's maximum heart rate. Each exercise session will consist of three phases; five-minutes warming up phase in form of stretching exercises and walking on the treadmill at the slowest speed, 20-minutes conditioning phase in form of walking on the treadmill at 50% of participants' maximum heart rate in the first two weeks then progressed gradually to reach the 70% of maximum heart rate by the 12th weeks", and five-minutes cool down phase that will be constant as warming up phase. During the training, the patient's blood pressure, heart rate, and breathing pattern will be frequently monitored . Also, the will be asked to follow a diet protocol designed by the nutrition specialist that rich in in vitamin D, fibers, and multiple nuts and seeds such as almond, walnut, pistachio, sunflower seeds, flax seeds and sesame seed to improve immune system for 12 weeks.

Group B (Aerobic training group): Patients will practice the aerobic training only like that of group A for 30 minutes, three sessions per week for 12 weeks.

Group C (Diet protocol group): Patients will only follow the same diet protocol that will be prescribed to group A for 12 weeks All patients in all groups will receive the same medical and traditional physical therapy in form of proper positioning and splinting and stretching, RoM, graduated strengthening exercises.

ELIGIBILITY:
Inclusion Criteria:

* Patients from both genders.
* The age ranges from 25 to 40 years.
* Weight range 60-85 kg, height 155- 170 cm.
* Total burned surface area (TBSA) was 20- 40% measured by the rule of nines.
* Thermal burn.
* Burn depth, partial-thickness burn injury.
* Patient will participate in the study one month after discharge.

Exclusion Criteria:

* Inhalation injury.
* Leg amputation.
* Any limitation in LL range of motion.
* Auditory or visual problems.
* Congenital musculoskeletal deformities, especially in the foot.
* Psychiatric disorders.
* Paralysis.
* Cardiac abnormalities or cardiac pacemakers.
* Patients who participated in any rehabilitation program before the study that may affect our results.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2024-02-19 (Estimated); Study Completion 2024-05-19 (Estimated)

PRIMARY OUTCOMES:
The immune markers | Three months
  total lymphocyte count (TLC) in 10^9 cells/liter will be measured
Neutrophil to lymphocyte ratio (NLR) | Three months
  The immune markers
Platelet to lymphocyte ratio (PLR) | Three months
  The immune markers

SECONDARY OUTCOMES:
The Arabic version of post traumatic stress disorder PTSD Checklist Civilian Version | Three months
  It is a 17-item self-report scale that measures PTSD symptom severity
The quality of life (QoL) | Three months
  Burn Specific Health Scale-Brief (BSHS-B) questionnaire will be used for the assessment of general, physical, mental, and social health aspects of the burn survivors

CONTACTS AND LOCATIONS:
Overall Officials: A G Elsayed, PHD, Study Chair — Cairo University
Locations (1):
- Faculty of Physical therapy, Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No